CLINICAL TRIAL: NCT01215344
Title: Impact of First Autologous Transplant on Minimal Residual Disease Markers in Previously Untreated Myeloma Undergoing Initial Treatment With Velcade Based Therapy
Brief Title: First Autologous Transplant on Minimal Residual Disease Markers in Previously Untreated Myeloma Undergoing Initial Treatment With Velcade
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Responsible Party: Principal Investigator, Madan Jagasia, MD, Associate Professor of Medicine; Director, Outpatient Transplant Program; Section Chief, Hematology and Stem Cell Transplant; Hematologist/Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VICC BMT 1020
Record Dates: First submitted 2010-10-04; First posted 2010-10-06 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2018-04

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Lenalidomide; Dexamethasone; Diphosphonates; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VRD (Experimental): VELCADE, Lenalidomide, Dexamethasone
  Interventions: Drug: VELCADE; Drug: Lenalidomide; Drug: Dexamethasone; Drug: DVT prophylaxis; Drug: Bisphosphonates
- VDD (Experimental): VELCADE, liposomal doxorubicin, dexamethasone
  Interventions: Drug: VELCADE; Drug: DVT prophylaxis; Drug: Liposomal doxorubicin; Drug: Dexamethasone

INTERVENTIONS:
Drug: VELCADE — 1.3 mg/m2 by IV on days 1, 4, 8, 11 of each cycle
Drug: Lenalidomide — 25 mg by mouth on days 1-4 of each cycle
  Arms: VRD
Drug: Dexamethasone — 20 mg the day before and the day after receiving VELCADE
  Arms: VRD
Drug: DVT prophylaxis — At least one asprin 81 mg per day. Other option per physician's choice
Drug: Bisphosphonates — Zoledronic acid by IB or pamidronate by IV can be used as per standard of care.
  Arms: VRD
Drug: Liposomal doxorubicin — 30 mg/m2 on day 4 of each cycle
  Arms: VDD
Drug: Dexamethasone — 40 mg by mouth on days 1-4, 8-11, and 15-18 of cycle 1 and days 1-4 on cycle 2-4
  Arms: VDD

SUMMARY:
The purpose of this study is to study the MRD status after VELCADE based induction therapy (VELCADE, lenalidomide, dexamethasone or VELCADE, liposomal doxorubicin, dexamethasone) in patients with previously untreated multiple myeloma and study the impact of HDC and ASCT on MRD status post-transplant. Our hypothesis is that MRD-status will continue to increase significantly at 3 months post-transplant and will validate that HDC and ASCT needs to be performed even when patients have achieved major response after induction therapy with novel agents.

ELIGIBILITY:
Inclusion Criteria:

Confirmed Multiple Myeloma as defined below within 120 days of starting cycle 1:

* Bone marrow plasmacytosis with ≥ 10% plasma cells or sheets of plasma cells or biopsy proven plasmacytoma
* Presence of M protein in serum or urine or both. Conventional M spike, serum free light chains, or 24 hour urine study. Non-secretory myeloma is not eligible for this study.
* In addition patient must have one of the following organ dysfunction criteria
* Hypercalcemia
* Renal insufficiency
* Anemia
* Bone disease manifested by lytic lesion or osteoporosis (if osteoporosis is the only organ dysfunction criteria then BM should have ≥ 30% plasma cells)
* Confirmed Multiple myeloma as defined above within 90 days of starting cycle 1
* The following study assessments must be fulfilled and must be obtained with four weeks of starting cycle 1
* Hemoglobin > 7 g/dL, Platelet count > 75 X 10 to 9th power/L, and Absolute neutrophil count > 1 X 10 to 9th power/L
* Creatinine <2.5 mg/dL or calculated creatinine clearance > 30 ml/min/1.72 m2
* Bilirubin ≤ 1.5 mg/dL X ULN
* SGPT (ALT) and SGOT (AST) ≤ 2.5 times the upper limit of normal
* Ejection fraction ≥ 45% as measured by a MUGA scan or 2 D echocardiogram
* Pulmonary function tests show >60% predicted values for FVC, FEV1, and DLCO FEV1 must be > 1 liter.
* No prior systemic therapy with the exception of bisphosphonates for MM
* Prior glucocorticoid therapy for the treatment of multiple myeloma is not permitted EXCEPT if used in conjunction with palliative radiation to prevent vasogenic edema. In that case steroids should have been used for less than 7 days. Prior steroid use for non-malignant disorders is permitted and should have been restricted to less than the equivalent of prednisone 10 mg per day. Prior or concurrent topical or localized steroid therapy to treat non-malignant disorders is permitted
* Prior palliative and/ or localized radiation therapy is permitted provided at least 4 weeks have passed from date of last radiation therapy to starting cycle 1.
* Patients with prior solitary plasmacytoma treated with radiation therapy with curative intent are eligible if the disease has now progressed to active multiple myeloma and meeting all eligibility criteria for the protocol
* ECOG PS 0, 1 or 2
* For women of childbearing potential a negative serum pregnancy test is required within 4 weeks of starting cycle 1 and then every 4 weeks during the first 4 cycles of induction therapy
* Women of child bearing potential must be willing to refrain from sexual intercourse or willing to employ a dual method of contraception, one of which is highly effective (IUD, birth control pills, tubal ligation or partner's vasectomy) and another additional method (condom, diaphragm, or cervical cap) during the entire course of the study (start of therapy until 30 days after stem cell transplant).
* Sexually active males should be willing to use a condom (even if they have had a prior vasectomy) while having intercourse with any women during the course of the study (start of therapy until 30 days after stem cell transplant).
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

Exclusion Criteria:

* Patients with smoldering myeloma or monoclonal gammopathy of unknown significance are not eligible
* Age > 70 years or < 18 years is not eligible
* Patient has > 1.5 × ULN Total Bilirubin
* Grade 2 or higher peripheral neuropathy due to ANY cause
* High index of suspicion of primary amyloid light chain (AL) amyloidosis.
* Patients with uncontrolled inter-current illness including uncontrolled hypertension, symptomatic congestive heart failure, unstable angina, uncontrolled cardiac arrhythmia, uncontrolled psychiatric illness or social situation that would limit compliance or a prior history of Steven Johnson syndrome
* Patients must not have a history of current or previous deep vein thrombosis or pulmonary embolism regardless of whether or not the patient is receiving anticoagulation therapy
* Female patients who are breastfeeding or pregnant.
* Patients known to be HIV positive
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure (see section 31.3), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
* Patient has hypersensitivity to VELCADE, boron or mannitol.
* Patient has received other investigational drugs within 14 days before enrollment
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-11; Primary Completion 2015-11 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madan Jagasia, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (2):
- United States (2):
  - University of Tennessee Cancer Institute, Boston Baskin Cancer Group, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

REFERENCES:
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://www.vicc.org/ct/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants participated in this trial at Vanderbilt-Ingram Cancer Center in Nashville, TN and the Boston Baskin Cancer Group in Memphis, TN. A total of 52 people consented to take part in this study and 15 were ineligible. One participant had disease progression before beginning treatment and wasn't assigned to a treatment arm.
Groups:
- VRD (VELCADE, Lenalidomide, Dexamethasone): VELCADE, Lenalidomide, Dexamethasone
  VELCADE: 1.3 mg/m2 by IV on days 1, 4, 8, 11 of each cycle
  Lenalidomide: 25 mg by mouth on days 1-4 of each cycle
  Dexamethasone: 20 mg the day before and the day after receiving VELCADE
  DVT prophylaxis: At least one asprin 81 mg per day. Other option per physician's choice
  Bisphosphonates: Zoledronic acid by IB or pamidronate by IV can be used as per standard of care.
- VDD (VELCADE, Liposomal Doxorubicin, Dexamethasone): VELCADE, liposomal doxorubicin, dexamethasone
  VELCADE: 1.3 mg/m2 by IV on days 1, 4, 8, 11 of each cycle
  DVT prophylaxis: At least one asprin 81 mg per day. Other option per physician's choice
  Liposomal doxorubicin: 30 mg/m2 on day 4 of each cycle
  Dexamethasone: 40 mg by mouth on days 1-4, 8-11, and 15-18 of cycle 1 and days 1-4 on cycle 2-4
Period: Overall Study
Arm/Group | VRD (VELCADE, Lenalidomide, Dexamethasone) | VDD (VELCADE, Liposomal Doxorubicin, Dexamethasone)
Started | 33 | 3
Completed | 23 | 3
Not Completed | 10 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VRD (VELCADE, Lenalidomide, Dexamethasone) | VDD (VELCADE, Liposomal Doxorubicin, Dexamethasone) | Total
Number analyzed (Participants) | 33 | 3 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 3 | 27
  >=65 years | 9 | 0 | 9
Age, Continuous [Median (Standard Deviation); unit: years] | 60 (8.71411) | 48 (4.642796) | 58.5 (8.803890)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 0 | 13
  Male | 20 | 3 | 23
Region of Enrollment [Number; unit: participants]
  United States | 33 | 3 | 36

OUTCOME MEASURES:

1. Primary Outcome: The Percent of Patients With Minimal Residual Disease (MRD) Status Changing to Negative at Day 100 (Post-AHCT), Among Patients With MRD Positive at the End of Induction (EOI).
Description: Patients were treated with induction therapy (VRD) followed by autologous hematopoietic cell transplant (AHCT). MRD status of a patient with at least partial response was evaluated at the end of induction (EOI) and day 100 (post-AHCT). MRD of a patient is measured by seven-color flow cytometry.
Time Frame: 6-months post ASCT
Population: Newly diagnosed, symptomatic multiple myeloma (MM) patients. Patients were treated with induction therapy VRD followed by AHCT. MRD staus was evaluated for patients with at least partial response at the end of induction (EOI) therapy. Ten of these patients had MRD negative at EOI.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- VELCADE, Lenalidomide, Dexamethasone (VRD): VELCADE, Lenalidomide, Dexamethasone
  VELCADE: 1.3 mg/m2 by IV on days 1, 4, 8, 11 of each cycle
  Lenalidomide: 25 mg by mouth on days 1-4 of each cycle
  Dexamethasone: 20 mg the day before and the day after receiving VELCADE
  DVT prophylaxis: At least one asprin 81 mg per day. Other option per physician's choice
  Bisphosphonates: Zoledronic acid by IB or pamidronate by IV can be used as per standard of care.
- VELCADE, Liposomal Doxorubicin, Dexamethasone (VDD): VELCADE, liposomal doxorubicin, dexamethasone
  VELCADE: 1.3 mg/m2 by IV on days 1, 4, 8, 11 of each cycle
  DVT prophylaxis: At least one asprin 81 mg per day. Other option per physician's choice
  Liposomal doxorubicin: 30 mg/m2 on day 4 of each cycle
  Dexamethasone: 40 mg by mouth on days 1-4, 8-11, and 15-18 of cycle 1 and days 1-4 on cycle 2-4
Arm/Group | VELCADE, Lenalidomide, Dexamethasone (VRD) | VELCADE, Liposomal Doxorubicin, Dexamethasone (VDD)
Number analyzed (Participants) | 20 | 0
percentage of participants | 30 [11 to 60] |

2. Secondary Outcome: Progression Free Survival by MRD Status at Day 100.
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: up to 7 years
Population: Patients with MRD status information at the EOI and day 100 (post-AHCT).
Measure: Median (95% Confidence Interval); unit: years
Groups:
- MRD Negative at Day 100: Patients with MRD status negative at day 100 (post-AHCT). They have MRD negative or positve at EOI.
- MRD Status Positive at Day 100 (Post-AHCT): Patients with MRD status stay positive at both EOI and day 100.
Arm/Group | MRD Negative at Day 100 | MRD Status Positive at Day 100 (Post-AHCT)
Number analyzed (Participants) | 13 | 7
years | 2.64 [0.73 to NA] — The value is not estimable. | NA [NA to NA] — These values are not estimable because no event happened yet.

ADVERSE EVENTS:
Arm/Group | VRD (VELCADE, Lenalidomide, Dexamethasone) | VDD (VELCADE, Liposomal Doxorubicin, Dexamethasone)
Serious Adverse Events (participants affected / at risk) | 9/33 | 0/3
Other Adverse Events (participants affected / at risk) | 31/33 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VRD (VELCADE, Lenalidomide, Dexamethasone) (N=33) | VDD (VELCADE, Liposomal Doxorubicin, Dexamethasone) (N=3)
Decreased hemoglobin (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Infection with normal ANC - Esophagus (Infections and infestations) | 1 (1) | 0 (0)
dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Potassium low (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gastric Schwannoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
GI bleed (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Elevated creatinine (Investigations) | 1 (1) | 0 (0)
Hip fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Rash, desquamation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VRD (VELCADE, Lenalidomide, Dexamethasone) (N=33) | VDD (VELCADE, Liposomal Doxorubicin, Dexamethasone) (N=3)
Nausea (Gastrointestinal disorders) | 14 (21) | 1 (2)
Constipation (Gastrointestinal disorders) | 12 (15) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 9 (12) | 0 (0)
Mucositis/stomatitis (Gastrointestinal disorders) | 7 (7) | 3 (3)
Anorexia (Gastrointestinal disorders) | 5 (6) | 0 (0)
Vomiting (General disorders) | 5 (6) | 0 (0)
Gastritis (Gastrointestinal disorders) | 3 (4) | 0 (0)
Heartburn (Gastrointestinal disorders) | 2 (5) | 0 (0)
Taste alteration (Gastrointestinal disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 15 (21) | 3 (5)
Fever (General disorders) | 8 (8) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (2)
Weight gain (Investigations) | 2 (2) | 0 (0)
Weight loss (Investigations) | 2 (7) | 0 (0)
Neuropathy: sensory (Nervous system disorders) | 16 (31) | 2 (4)
Dizziness (Nervous system disorders) | 5 (8) | 0 (0)
Depression (Psychiatric disorders) | 3 (4) | 0 (0)
Neuropathy (motor) (Nervous system disorders) | 3 (4) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
Gastrointestinal (other) (Gastrointestinal disorders) | 7 (9) | 0 (0)
Neurological (other) (Nervous system disorders) | 5 (6) | 0 (0)
Pain (other) (General disorders) | 10 (12) | 0 (0)
Headache (Nervous system disorders) | 5 (9) | 1 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Muscle pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Pain-chest wall (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
neuralgia/peripheral nerve (Nervous system disorders) | 2 (3) | 0 (0)
Throat pain (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Metabolic/Laboratory (other) (Investigations) | 4 (5) | 1 (5)
Potassium, serum-low (Metabolism and nutrition disorders) | 5 (5) | 0 (0)
Glucose high (Metabolism and nutrition disorders) | 2 (2) | 2 (6)
Calcium low (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Alkaline phosphatase (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 7 (11) | 1 (3)
Skin, other (Skin and subcutaneous tissue disorders) | 5 (9) | 0 (0)
Itching (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash, erythema multiforme (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash on hand-foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Muscle/soft tissue, other (Musculoskeletal and connective tissue disorders) | 8 (18) | 0 (0)
Gait disturbance (General disorders) | 3 (3) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5) | 0 (0)
Infection, other (Infections and infestations) | 2 (2) | 0 (0)
Infection with normal ANC - skin (cellulitis) (Infections and infestations) | 2 (2) | 0 (0)
Infection with normal ANC - Upper airway NOS (Infections and infestations) | 2 (2) | 0 (0)
Infection with normal ANC - Eye NOS (Infections and infestations) | 2 (2) | 0 (0)
Infection with normal ANC - Abdomen NOS (Infections and infestations) | 0 (0) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 9 (16) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Upper Respiratory - other (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Sinus reactions (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Voice change (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Neutrophils/granulocytes (Investigations) | 6 (10) | 1 (2)
Hemoglobin (Blood and lymphatic system disorders) | 5 (8) | 1 (2)
Platelets (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Leukocytes (Blood and lymphatic system disorders) | 3 (6) | 0 (0)
Blood/bone marrow - other (Blood and lymphatic system disorders) | 2 (4) | 0 (0)
Swelling of limb (General disorders) | 7 (10) | 0 (0)
Lymphatics - other (Blood and lymphatic system disorders) | 3 (4) | 0 (0)
Hypetension (Vascular disorders) | 4 (7) | 1 (1)
Cardiac (other) (Cardiac disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 2 (2)
Autoimmune reaction (Immune system disorders) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 3 (3) | 0 (0)
Renal (other) (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 2 (2) | 0 (0)
Flu-like syndrome (General disorders) | 3 (3) | 0 (0)
Low thyroid function (Endocrine disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes